CLINICAL TRIAL: NCT01135810
Title: Resting State Functional MRI Investigation of Hypnotic Trance and Mindfulness Meditation
Brief Title: Functional Magnetic Resonance Imaging (MRI) of Hypnosis and Mindfulness Meditation
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Jak, Lulu Sam Willson Professor, Stanford University
Other Study IDs: SU-05252010-6143; 17562
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Hypnosis
Keywords: healthy subjects
MeSH Terms: interventions — Hypnosis; Meditation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Hypnosis
Behavioral: Meditation

SUMMARY:
Hypnotic trance and mindfulness meditation have both been shown to have benefits for physical health. The current study seeks to determine if there are distinct patterns of brain activity that correlate with hypnotic trance, mindfulness meditation or both, and to relate these patterns to measurable markers of physical well-being. Precise neuroimaging of heightened attentional states will guide future researchers and practitioners toward more effective techniques of mind/body control.

DETAILED DESCRIPTION:
Our goal is to determine the functional brain networks that define and distinguish two induced states of sustained attention -- hypnosis and mindfulness -- that may be of substantial relevance to medicine.

Defining the neural underpinnings of these states would have broad implications for understanding how cognitive states emerge from functional networks, how they affect peripheral autonomic nervous system activity, and how their therapeutic efficacy can be optimized.

We propose a functional MRI study using resting state methodology to study 20-40 subjects from each of the four following groups:

1. Highly hypnotizable subjects
2. Minimally hypnotizable subjects
3. Experienced mindfulness meditators
4. Novice mindfulness meditators. The ability to be hypnotized is a stable and measurable trait that can be pre-screened and quantified. Dr. Spiegel will select subjects according to their ability to be hypnotized prior to the MRI visit (see ?recruiting? below). We will seek greatest contrast between groups by enrolling those with the highest (8-10) and lowest (0-2) scores on the Hypnotic Induction Profile. The presence of a poorly hypnotizable group allows for a control condition of those who have undergone an identical induction routine without achieving hypnotic trance. Similarly, novice meditators will serve as a control for the group experienced in mindfulness meditation.

Prior studies have shown differences in both brain activation and grey matter volume associated with longer practice of meditation (> 4 years) compared with novice meditators. As such, experienced meditators will be defined as those with a regular meditation practice of four years or longer. Novice meditators will be new practitioners who are interested in mindfulness meditation practice, and who completed a one-hour meditation training during the week before their study participation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not have contraindications to the MRI exam, such as metal in the body.

Exclusion Criteria:

* Contraindications to the MRI exam, such as metal in the body.
* Use of psychotropic medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects who score in diverse ranges on hypnotic induction profiles or who are experienced Mindfulness Meditators.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
MRI scan: brain activity | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States